CLINICAL TRIAL: NCT03614715
Title: Comparative Trial of the Pharmacokinetics and Pharmacodynamics of Intramuscularly Injected CinnoVex® and Avonex® in Healthy Volunteers
Brief Title: Pharmacokinetics and Pharmacodynamics of CinnoVex (Interferon Beta-1a) Compared to Avonex (Interferon Beta-1a)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MC-CINNA-PKPD-01; 2016-000139-41 (EudraCT Number)
Record Dates: First submitted 2018-07-14; First posted 2018-08-03 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2018-07

CONDITIONS: Bioequivalence; Healthy
MeSH Terms: interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CinnaGen interferon beta-1a (Experimental): CinnoVex® (IFNβ-1a, Prefilled syringe produced by CinnaGen Company) in prefilled syringe in healthy volunteers. (Stage 1: 30 µg or 60 µg)(Stage 2: 30 µg)
  Interventions: Drug: Interferon Beta-1A
- Biogen interferon beta-1a (Active Comparator): Avonex® (IFNβ-1a, Prefilled syringe produced by Biogen Company) in prefilled syringe in healthy volunteers. (Stage 1: 30 µg or 60 µg)(Stage 2: 30 µg)
  Interventions: Drug: Interferon Beta-1A

INTERVENTIONS:
Drug: Interferon Beta-1A — A single dose of Interferon Beta-1A (Stage 1: 30 or 60 µg, stage 2: 30 µg) was administered IM to healthy subjects (cross over treatment)
  Other Names: CinnoVex; Avonex

SUMMARY:
The primary objective of the trial is to investigate the biosimilarity of CinnoVex® by comparing its pharmacokinetics (PK) and pharmacodynamics (PD) to its originator, Avonex®, in a crossover manner in healthy female and male volunteers after administration of a single dose of 30 µg or 60 µg of Interferon beta-1a.

The secondary objectives of the study are:

* To further compare the PK of CinnoVex® and Avonex®.
* To further compare the PD of CinnoVex® and Avonex®.
* To assess the safety of CinnoVex®.

DETAILED DESCRIPTION:
This trial will be a double-blind, randomised, active-controlled, single-centre, two-stage crossover trial with administration of single doses of CinnoVex® and Avonex®. Stage 1 includes comparison of 30 µg and 60 µg IM doses in 16 healthy volunteers (eight subjects on each dose level, each subject will be administered one dose of each product as 30 µg or 60 µg doses in a crossover manner and in randomised order). After interim analysis of the PK and PD results of these 16 subjects and evaluation of the data by an expert data monitoring committee (DMC), Stage 2 will investigate the selected dose. The sample size of Stage 2 will be determined in the interim analysis so that a sufficient number of additional healthy volunteers are added to one or both dose levels to ensure adequate statistical power for the study's objectives, to evaluate biosimilarity. Up to 48 additional healthy volunteers may be added at this stage.

Subjects will undergo screening assessments before their first treatment visit. A total of 16 healthy volunteers will be selected for Stage 1 and 24 or 48 will be selected for Stage 2 according to the inclusion and exclusion criteria. To reveal possible differences in the trial outcomes between the sexes, approximately equal numbers of male and female subjects will be included. The trial will be performed in healthy adult volunteers with a maximum age of 45 years, to limit variability that may result from including older adults.

Eligibility of subjects will be confirmed prior to each IMP administration with a pregnancy test (female subjects with childbearing potential), a urine drug screen and an alcohol breath test. In addition, the subjects will be asked about current illnesses, subjective well-being, and concomitant medications. A physical examination will take place, if indicated.

The subjects will participate in 2 treatment periods in sequential order; treatment period 1 starts when the first IMP is administered and treatment period 2 starts when the second IMP is administered. The two treatment administrations of individual subjects will be separated by at least 14 days.

Blood samples will be collected prior to and at scheduled time points after the IMP administration. Plasma concentrations of IFNβ-1a and concentrations of the selected biomarkers in serum and blood will be determined. The total volume of blood collected from each subject during the trial is less than 500 ml.

Safety will be assessed by recording blood pressure (BP), heart rate (HR), body temperature and subjective symptoms at scheduled time points after IMP administration. AEs and concomitant medications will be recorded throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent (IC) to participate in the trial, to comply with the trial procedures, and to abide by the trial restrictions.
2. Be aged between 18 and 45 years with sufficient command of the Finnish language to be able to provide valid IC and to communicate adequately with the trial personnel.
3. Have a Body Mass Index (BMI) between 18 and 28 kg/m2.
4. Have good general health according to medical history, physical examination, ECG recording and clinical laboratory assessments.
5. Female subjects of child-bearing potential must agree to use a medically accepted method of contraception during the trial and one month after the end of the trial. Acceptable methods of contraception include the following:

   * Stable oral/transdermal/injectable hormonal contraceptive regimen without breakthrough uterine bleeding and condom/spermicide.
   * Intrauterine device (inserted at least 2 months prior to Screening visit) used with spermicide/condom.
   * Condom (male or female) with spermicide
   * Vasectomy of the male partner in conjunction with condom or spermicide.

Exclusion Criteria:

* 1) Be doubtful about his/her availability to complete the trial. 2) Have unsuitable veins for repeated venipuncture. 3) Be pregnant, or intend to become pregnant during the trial, or be lactating. 4) Have a history or evidence of clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic, endocrine, neurological, psychiatric or other major disease.

  5) Have any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug.

  6) Have strong susceptibility to allergic reactions or history of allergy to any of the components of the IMP.

  7) Have clinically significant illness within 4 weeks before the start of the trial.

  8) Have any abnormal laboratory value or physical finding which may interfere with the interpretation of the test results or cause a health hazard for the subject if he/she takes part in the trial.

  9) Have any condition requiring regular concomitant medication or use of any medication that might affect the trial results or cause a health hazard to the subject within 2 weeks prior to the start of the trial; hormonal contraception and hormone replacement therapy are allowed.

  10) Have history of alcohol abuse or drug addiction or a positive result in the urine drug screen or breath alcohol test, or report consumption of more than 14 units of alcohol per week on a regular basis (1 unit = 4 cl of spirits of equivalent).

  11) Have a history of smoking >10 cigarettes per day. 12) Participate in another drug trial or donation of blood within 90 days before first IMP administration in this trial.

  13) Have participated before in a clinical study investigating a Type I Interferon or have been treated with a Type I Interferon before.

  14) Be under anti-doping control. 15) Be at imminent risk of self-harm, based on clinical interview and responses on the Columbia Suicide Severity Rating Scale (C-SSRS), or of harm to others in the opinion of the investigator. Subjects must be excluded, if they report suicidal ideation with intent, with or without a plan or a method (e.g., positive response to items 4 or 5 in assessment of suicidal ideation on the C-SSRS) in the past two months or suicidal behaviour in the past six months.

  16) Have any other condition that in the opinion of the investigator would interfere with the evaluation of the trial results or constitute a health hazard for the subject.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
AUCt of IFNβ-1a | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  Area under the plasma concentration curve from the time of IMP administration to the last observed concentration at last time point t, calculated using the linear trapezoidal rule
Cmax of IFNβ-1a | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  Maximum concentration of IFNβ-1a in plasma

SECONDARY OUTCOMES:
tmax of IFNβ-1a | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  Time to maximum concentration of IFNβ-1a in plasma
t½ of IFNβ-1a | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  Elimination half-life of IFNβ-1a (if evaluable)
AUCinf of IFNβ-1a | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  Area under the concentration curve extrapolated to infinite time, if allowed by the concentration data (if Kel is evaluable)
VD | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  Volume of distribution
MRT | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  Mean residence time
CL | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  Clearance
AUC0-168 of neopterin | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  AUC0-168 of neopterin concentrations in serum
AUC0-168 of interleukin (IL)-10 | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  AUC0-168 of interleukin (IL)-10 concentrations in serum
AUC0-168 of IL-4 | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  AUC0-168 of IL-4 concentrations in serum
AUC0-168 of β2-microglobulin | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  AUC0-168 of β2-microglobulin concentrations in serum
AUC0-168 of MxA | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  AUC0-168 of MxA concentrations in whole blood
Concentrations of MxA in whole blood | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  validated ELISA methods
concentrations of neopterin in serum | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  validated ELISA methods
concentrations of β2-microglobulin in serum | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  validated ELISA methods
concentrations of IL-4 in serum. | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  validated ELISA methods
concentrations of IL-10 in serum | blood samples will be drawn prior to Investigational Medicinal Product administration, and then at the following times after dosing: 12, 14, 16, 18, and 24 hours, and mornings of Day 3, Day 4, Day 5, Day 6, and Day 8
  Validated ELISA methods
Adverse events | Prior to the Investigational Medicinal Product administration and up to 8 days after drug administration (cross over study)
  Recording from patients
Heart rate as vital signs | Prior to the Investigational Medicinal Product administration and up to 8 days after drug administration (cross over study)
  Record at CRF, changes will be presented using summary statistics
Body temperature as vital sign | Prior to the Investigational Medicinal Product administration and up to 8 days after drug administration (cross over study)
  Record at CRF, changes will be presented using summary statistics
ECG as vital sign | Prior to the Investigational Medicinal Product administration and up to 8 days after drug administration (cross over study)
  Record at CRF, changes will be presented using summary statistics
Supine blood pressure as vital sign | Prior to the Investigational Medicinal Product administration and up to 8 days after drug administration (cross over study)
  Record at CRF, changes will be presented using summary statistics

CONTACTS AND LOCATIONS:
Overall Officials: Mika Scheinin, MD, PhD, Principal Investigator — CRST, Itäinen Pitkäkatu 4B, FI-20520 Turku, Finland
Locations (1):
- CRST Oy, Clinical Research Services Turku Itäinen Pitkäkatu 4 B, 3rd floor, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lengyel P. Biochemistry of interferons and their actions. Annu Rev Biochem. 1982;51:251-82. doi: 10.1146/annurev.bi.51.070182.001343. No abstract available. PMID 6180680
- [Background] Pestka S, Langer JA, Zoon KC, Samuel CE. Interferons and their actions. Annu Rev Biochem. 1987;56:727-77. doi: 10.1146/annurev.bi.56.070187.003455. No abstract available. PMID 2441659
- [Background] Romano A, Sadan Y. Ten years of experience with human fibroblast interferon in treatment of viral ophthalmic infections. Metab Pediatr Syst Ophthalmol (1985). 1988;11(1-2):43-6. PMID 3076609
- [Background] Capalbo M, Palmisano L, Bonino F, Pellas C, Maset J. Intramuscular natural beta interferon in the treatment of chronic hepatitis B: a multicentre trial. Italian Hepatitis B Study Group. Ital J Gastroenterol. 1994 Jun;26(5):238-41. PMID 7919465
- [Background] Chemello L, Cavalletto L, Noventa F, Bonetti P, Casarin C, Bernardinello E, Pontisso P, Donada C, Casarin P, Belussi F, et al. Predictors of sustained response, relapse and no response in patients with chronic hepatitis C treated with interferon-alpha. J Viral Hepat. 1995;2(2):91-6. doi: 10.1111/j.1365-2893.1995.tb00012.x. PMID 7493303
- [Background] Miles SA, Wang HJ, Cortes E, Carden J, Marcus S, Mitsuyasu RT. Beta-interferon therapy in patients with poor-prognosis Kaposi sarcoma related to the acquired immunodeficiency syndrome (AIDS). A phase II trial with preliminary evidence of antiviral activity and low incidence of opportunistic infections. Ann Intern Med. 1990 Apr 15;112(8):582-9. doi: 10.7326/0003-4819-112-8-582. PMID 2109563
- [Background] Nagai M, Arai T. Clinical effect of interferon in malignant brain tumours. Neurosurg Rev. 1984;7(1):55-64. doi: 10.1007/BF01743290. PMID 6379511
- [Background] Placebo-controlled multicentre randomised trial of interferon beta-1b in treatment of secondary progressive multiple sclerosis. European Study Group on interferon beta-1b in secondary progressive MS. Lancet. 1998 Nov 7;352(9139):1491-7. PMID 9820296
- [Background] Hovanessian AG, Justesen J. The human 2'-5'oligoadenylate synthetase family: unique interferon-inducible enzymes catalyzing 2'-5' instead of 3'-5' phosphodiester bond formation. Biochimie. 2007 Jun-Jul;89(6-7):779-88. doi: 10.1016/j.biochi.2007.02.003. Epub 2007 Feb 20. PMID 17408844
- [Background] Scagnolari C, Duda P, Bagnato F, De Vito G, Alberelli A, Lavolpe V, Girardi E, Durastanti V, Trojano M, Kappos L, Antonelli G. Pharmacodynamics of interferon beta in multiple sclerosis patients with or without serum neutralizing antibodies. J Neurol. 2007 May;254(5):597-604. doi: 10.1007/s00415-006-0332-7. Epub 2007 Apr 10. PMID 17420930
- [Background] Casoni F, Merelli E, Bedin R, Sola P, Bertolotto A, Faglioni P. Is serum neopterin level a marker of responsiveness to interferon beta-1a therapy in multiple sclerosis? Acta Neurol Scand. 2004 Jan;109(1):61-5. doi: 10.1046/j.1600-0404.2003.00177.x. PMID 14653852
- [Background] Bertolotto A, Gilli F, Sala A, Audano L, Castello A, Magliola U, Melis F, Giordana MT. Evaluation of bioavailability of three types of IFNbeta in multiple sclerosis patients by a new quantitative-competitive-PCR method for MxA quantification. J Immunol Methods. 2001 Oct 1;256(1-2):141-52. doi: 10.1016/s0022-1759(01)00434-3. PMID 11516761
- [Background] Bertolotto A, Deisenhammer F, Gallo P, Solberg Sorensen P. Immunogenicity of interferon beta: differences among products. J Neurol. 2004 Jun;251 Suppl 2:II15-II24. doi: 10.1007/s00415-004-1204-7. PMID 15264108
- [Background] Williams GJ, Witt PL. Comparative study of the pharmacodynamic and pharmacologic effects of Betaseron and AVONEX. J Interferon Cytokine Res. 1998 Nov;18(11):967-75. doi: 10.1089/jir.1998.18.967. PMID 9858319
- [Background] Jacobs LD, Cookfair DL, Rudick RA, Herndon RM, Richert JR, Salazar AM, Fischer JS, Goodkin DE, Granger CV, Simon JH, Alam JJ, Bartoszak DM, Bourdette DN, Braiman J, Brownscheidle CM, Coats ME, Cohan SL, Dougherty DS, Kinkel RP, Mass MK, Munschauer FE 3rd, Priore RL, Pullicino PM, Scherokman BJ, Whitham RH, et al. Intramuscular interferon beta-1a for disease progression in relapsing multiple sclerosis. The Multiple Sclerosis Collaborative Research Group (MSCRG). Ann Neurol. 1996 Mar;39(3):285-94. doi: 10.1002/ana.410390304. PMID 8602746
- [Background] PRISMS Study Group and the University of British Columbia MS/MRI Analysis Group.. PRISMS-4: Long-term efficacy of interferon-beta-1a in relapsing MS. Neurology. 2001 Jun 26;56(12):1628-36. doi: 10.1212/wnl.56.12.1628. PMID 11425926
- [Background] Ben-Amor AF, Trochanov A, Fischer TZ. Cumulative Review of Thrombotic Microangiopathy, Thrombotic Thrombocytopenic Purpura, and Hemolytic Uremic Syndrome Reports with Subcutaneous Interferon beta-1a. Adv Ther. 2015 May;32(5):445-54. doi: 10.1007/s12325-015-0212-6. Epub 2015 May 20. PMID 25991578
- [Background] Munafo A, Trinchard-Lugan I I, Nguyen TX, Buraglio M. Comparative pharmacokinetics and pharmacodynamics of recombinant human interferon beta-1a after intramuscular and subcutaneous administration. Eur J Neurol. 1998 Mar;5(2):187-193. doi: 10.1046/j.1468-1331.1998.520187.x. PMID 10210831
- [Background] Di Girolamo G, Kauffman MA, Gonzalez E, Papouchado M, Ramirez A, Keller G, Carbonetto C, Dabsys S, Vidal A, Sterin-Prync A, Diez RA. Bioequivalence of two subcutaneous pharmaceutical products of interferon beta la. Arzneimittelforschung. 2008;58(4):193-8. doi: 10.1055/s-0031-1296492. PMID 18540482
- [Background] Malucchi S, Sala A, Gilli F, Bottero R, Di Sapio A, Capobianco M, Bertolotto A. Neutralizing antibodies reduce the efficacy of betaIFN during treatment of multiple sclerosis. Neurology. 2004 Jun 8;62(11):2031-7. doi: 10.1212/01.wnl.0000129265.73259.9e. PMID 15184610